CLINICAL TRIAL: NCT06665958
Title: Comparison of the Bioavailability of the Flavanol of Grape Extracts Administered in Capsule or in Gummy: a 4-way Randomized Crossover Study in Healthy Participants
Brief Title: Comparison of the Bioavailability of the Flavanol of Grape Extracts
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REC/24/0047
Record Dates: First submitted 2024-10-24; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Healthy Nutrition
Keywords: Flavan-3-ols, grape seed extracts; microbial metabolites; bioavailability; Flavan-3-ols; grape seed extracts
MeSH Terms: interventions — Polyphenols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: Polyphenol extract low dose (hard capsule) (Experimental): <2% flavanol monomer hard capsule
  Interventions: Dietary Supplement: Polyphenol extract
- Experimental: Polyphenol extract medium dose (hard capsule) (Experimental): 15% flavanol monomer hard capsule
  Interventions: Dietary Supplement: Polyphenol extract
- Experimental: Polyphenol extract medium dose (gummy) (Experimental): 15% flavanol monomer x2 gummy
  Interventions: Dietary Supplement: Polyphenol extract
- Experimental: Polyphenol extract high dose (hard capsule) (Experimental): 26% flavanol monomer hard capsule
  Interventions: Dietary Supplement: Polyphenol extract

INTERVENTIONS:
Dietary Supplement: Polyphenol extract — Single dose

SUMMARY:
Polyphenols are a group of naturally occurring compounds found in cocoa, teas, and grape seed extracts (GSE) that have been linked to various health benefits. This study will provide a greater insight into the relationship between polyphenol consumption and health, and could be used to help with the development of functional food products and novel supplements. Although the advantages of a polyphenol-rich diet are well-established, the bioavailability of GSE (a source of polyphenols) in the context of human digestion and beneficial properties are poorly understood.

The investigators will conduct an open-label, randomized, 4-way crossover design with the aim to explore the bioavailability of GSE-derived flavan-3-ols from GSE and their related microbial metabolites and advance understanding of the bioactive properties of flavan-3-ols contributing to the development of more effective dietary strategies and functional food products.

DETAILED DESCRIPTION:
(Poly)phenols a complex class of naturally occurring compounds have garnered increasing attention due to their putative bioactive effects. Flavan-3-ols a subgroup of polyphenols, predominantly found in cocoa, various teas (including black and green tea), and grape seed extracts (GSE), have been associated with various health benefits including cardioprotective, neuroprotective, and anti-inflammatory effects. Moreover, their monomeric forms catechin and epicatechin have been increasingly investigated for their antioxidant properties, which may contribute to the prevention of chronic diseases such as cardiovascular disorders, diabetes, and neurodegenerative conditions. Increasing number of large-scale intervention trials have reported an inverse correlation between a flavan-3-ol intake in range of 400 - 800 mg/d and the risk of cardiovascular disease. A finding that has been supported by the recent COSMOS trial which included >20,000 participants who consumed 600 mg/d, reporting a significant 15% reduction in total CVD events when compared to the placebo group.

Despite these benefits, the efficacy of flavan-3-ols is heavily dependent on their bioavailability. However, this is severely influenced by various factors including the chemical structure, dosage, and the food matrix. Moreover, after ingestion, very few (poly)phenols are readily absorbed within the small intestine and subsequently not present in the circulation as the parent compound but as simpler phenolics, derived from the colonic fermentation within the large intestine where they are metabolised by the local microbiota through a series of chemical modifications such as ring fission, and cleavage of ester and/or glycosidic bonds. The newly formed simple phenolics may then undergo a various transformations mediated in part by local epithelial cell producing phase I/II metabolites such as, phenyl-y-valerolactones (PVLs) and their related phenylvaleric acids (PVAs), indicating that it is these secondary metabolites that offer the described benefits post-absorption. Although these metabolites are thought to play significant roles in health outcomes, their identification and quantification remains a challenge due to the lack of reference standards in biological fluids. Moreover, the metabolic fate of these compounds is characterized by a high degree of inter-individual variability, which is further complicated by factors such as enterohepatic recirculation and the diverse metabolic capabilities of the gut microbiota. Research has demonstrated that encapsulation technologies can influence the bioavailability of polyphenols, with different delivery systems such as hard capsules and soft gummies affecting the dissolution rates and systemic exposure of these bioactive compounds. Given these complexities, there is an increasing need to further elucidate the pharmacokinetic profiles of flavan-3-ols and their metabolites to optimize their health benefits. To this end, the investigators seek to conduct an open-label, randomized, 4-way crossover design with the aim to explore the bioavailability of GSE-derived flavan-3-ols from GSE and their related microbial metabolites and advance understanding of the bioactive properties of flavan-3-ols contributing to the development of more effective dietary strategies and functional food products.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Aged 18-40 years at recruitment
* BMI ≥ 20 and < 30kg/m2
* Considered healthy based on their medical history and physical examination.
* Subjects capable of and willing to comply with the protocol and to give their written informed consent.

Exclusion Criteria:

* Existing chronic disease including any; cardiovascular, neurological, gastric/intestinal, hepatic/pancreatic, renal or hematological diseases, obstructive cardiomyopathy, myocardial infarction, intracranial hypertension, diabetes mellitus (type I or II), chronic kidney disease, clinically significant arrhythmia, metabolic anomaly, ischaemia heart disease.
* Uncontrolled Hypertension (>160/100 mm Hg) or hypotension (<100/60mm Hg)
* Current use of any medication or narcotics within 2 weeks prior to study entry.
* Currently on a clinically prescribed diet regimen.
* Self-reported alcohol intake of >10 units/ week
* Have taken antibiotic therapy within the last 3 months
* Following any specific diet (vegetarian, vegan, etc.)
* Consumption of dietary supplement(s) currently or within 4 weeks prior to study entry (i.e. botanicals, vitamins, minerals, amino acids).
* Weight change > 10% of total body weight within the 6 months before entry to study.
* Any intolerance or allergy documented or suspected to one of the components of the study products.
* Having a psychological or linguistic inability to sign the informed consent; Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision;
* Subject participating in another biomedical study or participation in another study within the 3 months before entry into this study.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological males
Enrollment: 25 (Estimated)
Dates: Start 2024-10-28 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration (µM) of flavan-3-ols monomer (poly)phenols. | Change over 24 hours compared across treatments
  Quantification by LC-MS/MS

SECONDARY OUTCOMES:
Plasma concentration (µM) of main flavan-3-ol metabolites. | Change over 24 hours compared across treatments
  Quantification by LC-MS/MS
Total excretion of primary flavanol metabolites (µM). | Change over 24 hours compared across treatments.
  Quantification by LC-MS/MS
Systolic Blood Pressure (mmHg) | Measured at 8 hours post-ingestion compared across treatments.
  Measured by branchial blood pressure monitor.
Diastolic Blood Pressure (mmHg) | Measured at 8 hours post-ingestion compared across treatments.
  Measured by branchial blood pressure monitor.

OTHER OUTCOMES:
Tolerance/Acceptability Questionnaire | Measured at 8 hours post-ingestion compared across treatments.
  Product appeal, gastrointestinal symptoms (e.g., stomachache, bloating, nausea) and willingness to continue consumption rated on a 4-point scale (1 = "least favorable" to 4 = "most favorable")

CONTACTS AND LOCATIONS:
Overall Officials: Chris Gill, Principal Investigator — Ulster University
Locations (1):
- Ulster University,Human Intervention Studies UnitColeraine, Co. Londonderry BT521SA, Coleraine, Co. Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No